CLINICAL TRIAL: NCT04838925
Title: Using Mobile Devices for Neurofeedback to Reduce Opioid Use in Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CrossComm, Inc. (Industry)
Collaborators: Duke University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00106634; 1R41DA053011-01 (NIH)
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pain; Opioid Use
Keywords: Chronic Pain; Opioids; Prescription Opioids; Pain; Musculoskeletal Pain; Mobile Apps; Mobile Health; Neurofeedback; EEG Feedback; Biofeedback; Alternative Therapy
MeSH Terms: conditions — Chronic Pain; Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Mobile Neurofeedback (Experimental): Participants engage in the use of a mobile neurofeedback intervention, which involves using a mobile app paired with an EEG headset, to achieve a calm, relaxed state. Participants will be instructed to use the intervention at a minimum of 10 minutes a day, 4 times a week for a total of 12 weeks.
  Interventions: Device: Mobile Neurofeedback App

INTERVENTIONS:
Device: Mobile Neurofeedback App — Neurofeedback intervention delivered via mobile app. Participants wear an EEG headset which is connected to a mobile app that delivers feedback about brainwave data indicating whether they are in a calm, relaxed state. Participants hear a lower/simple sound when they are below a target level and higher/richer sound when they approach or achieve their target.

SUMMARY:
The purpose of this study is to develop and test the feasibility of a commercially-ready mobile neurofeedback app for individuals with chronic pain. Thirty (30) participants who are prescribed opioids for chronic pain will use the new mobile neurofeedback app and an EEG headset for 10 minutes at a time, 4 times a week for 12 weeks and provide feedback about using the app.

DETAILED DESCRIPTION:
In this STTR Phase I project, CrossComm will collaborate with Duke University to develop a commercial-ready mobile neurofeedback technology and test its feasibility among patients using opioids to treat chronic pain. Specific Aim 1 is to develop a commercial-ready mobile neurofeedback app and will be built according to commercial standards of robustness and maintainability. Specific Aim 2 is to test feasibility of the commercially available mobile app in N=30 patients with chronic pain prescribed opioids. Participants will be recruited for a baseline interview with the Duke Behavioral Health & Technology Lab after passing a preliminary telephone screen. After providing informed consent, participants will provide data on demographics, pain symptoms, and opioid consumption. Each participant will download the mobile neurofeedback app to their smartphone and be instructed to use the intervention for 10 minutes a day, 4 times a week for 12 weeks. Study coordinators will conduct four teleconference sessions (weeks 1, 3, 6 and 9) to reinforce training, troubleshoot difficulties, and support intervention utilization. After the 12-week mobile neurofeedback intervention, the investigators will collect follow-up data, including pain measures, mobile app (usage, satisfaction, & usability), and user feedback on the human-computer interface. Data from these will inform further app refinement preparing for STTR Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Reports chronic pain (≥4 on 0-10 Numeric Rating Scale (NRS) on most days during the past 3 months)
* Prescribed opioids for pain management

Exclusion Criteria:

* History of seizures
* Plans to have pain-related surgery in the next 3 months
* Has an implanted medical device that could experience interference during EEG, such as a spinal cord stimulator or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Mobile App Usage | 12 weeks
  Objective data on number of mobile neurofeedback sessions completed by participants. Intervention adherence data will inform the feasibility of real-world use of the commercial-ready mobile app.

SECONDARY OUTCOMES:
Mobile App Satisfaction assessed on a 5-point Likert scale (1: very dissatisfied - 5: very satisfied) | At 3 month follow-up (end of intervention)
  Rating on a 5-point Likert scale (1: very dissatisfied - 5: very satisfied) of how satisfied participants were with the mobile neurofeedback app.
Mobile App Usability assessed by the System Usability Scale | At 3 month follow-up (end of intervention)
  The participant indicates level of agreement with 10 statements (1: strongly disagree - 5 strongly agree). Scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. (From: https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html) Higher scores indicate better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Elbogen, PhD, Principal Investigator — Duke University; Donald K Shin, Principal Investigator — CrossComm, Inc.
Locations (1):
- Duke University School of Medicine Department of Psychiatry, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No